CLINICAL TRIAL: NCT00429754
Title: A Pharmacokinetic Evaluation of the Addition of Aprepitant to the Bleomycin -Etoposide - Cisplatin (BEP) Treatment of Patients With Testis Carcinoma (A-BEP)
Brief Title: Pharmacokinetic Study of Aprepitant in BEP Treatment of Patients With Testis Carcinoma (A-BEP)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: change of study population and chemotherapeutic regimen
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF 06.01
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Nausea; Vomiting
Keywords: Nausea and vomiting after using cytostatic drugs
MeSH Terms: conditions — Nausea; Vomiting | interventions — Aprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aprepitant (Other): Aprepitant treatment
  Interventions: Drug: Aprepitant

INTERVENTIONS:
Drug: Aprepitant

SUMMARY:
The purpose of the study is to investigate whether there is an interaction occurs between etoposide and aprepitant in patients with testis carcinoma treated with the standard BEP regimen.

Also to determine how long treatment with aprepitant is necessary in BEP regimen for 5 consecutive days.

DETAILED DESCRIPTION:
Aprepitant is a novel, potent and selective nonpeptide neurokinin-1 receptor antagonist that was licensed in 2004 for the prevention of acute and delayed nausea and vomiting associated with highly emetogenic cancer chemotherapy.More recently the indication for use of aprepitant was extended to patients with moderately emetogenic chemotherapy. Based on experience with the use of aprepitant it appears rational to consider aprepitant as part of the anti-emetic regimen for patients treated with BEP. There are, however, no published data available for the use of aprepitant in this situation.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 75 years of age
* able and willing to sign Informed Consent Form
* subject has an indication for treatment with BEP regimen
* subject is expected to receive at least 2 cycles of BEP regimen
* subject is able to swallow capsules

Exclusion Criteria:

* documented history of sensitivity/idiosyncrasy to aprepitant or excipients
* relevant history or condition that might interfere with drug absorption
* history of or current abuse of drugs, alcohol or solvents
* inability to understand nature and extent of the trial and the procedures
* participation in a drug trial within 30 days prior to the first dose
* febrile illness within 3 days before the first dose
* use of agents that are known to interfere with aprepitant pharmacokinetics
* abnormal liver or renal function

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2008-09

PRIMARY OUTCOMES:
Pharmacokinetic blood samples will be taken at day 2 at pre-dose,
at 1/2 hour after intake, at 1, 4, 6, 8 and 24 hours (is day 3) after intake of medication.
Also at day 5 at the same time points blood samples will be taken.

SECONDARY OUTCOMES:
Nausea and vomiting questionnaires will be answered at day 1,2,3,4,5,6,8 en 15.

CONTACTS AND LOCATIONS:
Overall Officials: David M. Burger, PharmD PhD, Principal Investigator — Radboud University (RUNMC)